CLINICAL TRIAL: NCT04522843
Title: Analysis of Intestinal Defensin Expression in Patients With Acute Graft-versus-Host Disease (GVHD)
Brief Title: Analysis of Intestinal Defensin Expression in Acute GVHD
Status: Completed | Type: Observational
Sponsor: University of Freiburg (Other)
Responsible Party: Principal Investigator, Robert Zeiser, Director of the Division of Tumor Immunology, University of Freiburg
Other Study IDs: GVHD_Def
Record Dates: First submitted 2020-08-18; First posted 2020-08-21 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: GVHD,Acute; Ulcerative Colitis; Morbus Crohn
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Uninflamed intestine: Patients who underwent diagnostic endoscopy and received a diagnosis of no intestinal inflammation
- Colitis: Patients with active colitis
- Acute GVHD: Patients with acute gastrointestinal (GI) GVHD

SUMMARY:
This study has the aim to analyze intestinal expression of endogenous antimicrobial peptides in patients with acute GVHD. The expression will be compared to intestinal expression of defensins in patients with colitis and patients without intestinal inflammation.

DETAILED DESCRIPTION:
Acute graft-versus-host disease (GVHD) is a major cause of morbidity and mortality in patients undergoing allogeneic hematopoietic cell transplantation (allo-HCT). Acute GVHD is characterized by complex deficiencies of the mucosal antimicrobial barrier and intestinal dysbiosis, which contribute to disease pathogenesis. Defensins are endogenous epithelial cell-derived antimicrobial peptides, which can protect epithelial barrier integrity, shape the intestinal microbiota composition and contribute to host immunoregulation. Deregulated expression of defensins has been reported in patients with colitis, including Chron's Disease and ulcerative colitis.

In this study, the investigators aim to analyze the expression of defensins in the intestine of patients with acute GVHD to study whether it is deregulated. The results will be valuable to study the role of defensins during acute GVHD pathogenesis or as potential biomarkers for disease activity.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* diagnostic endoscopy was performed
* diagnosis results available
* written informed consent
* ability to understand the nature of the study and the study related procedures and to comply with them

Exclusion Criteria:

* age < 18 years
* gastrointestinal cancer
* lack of informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who underwent diagnostic endoscopy
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Defensin Expression (mRNA) | 3 years
  Analysis of alpha-defensin and beta-defensin mRNA expression by realtime PCR (qRT-PCR)
Defensin Expression (peptide) | 3 years
  Analysis of alpha-defensin and beta-defensin levels by immunohistochemistry

CONTACTS AND LOCATIONS:
Overall Officials: Robert Zeiser, Prof. Dr., Principal Investigator — Medical Center University of Freiburg
Locations (1):
- Medical Center University of Freiburg, Freiburg im Breisgau, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wehkamp J, Fellermann K, Herrlinger KR, Baxmann S, Schmidt K, Schwind B, Duchrow M, Wohlschlager C, Feller AC, Stange EF. Human beta-defensin 2 but not beta-defensin 1 is expressed preferentially in colonic mucosa of inflammatory bowel disease. Eur J Gastroenterol Hepatol. 2002 Jul;14(7):745-52. doi: 10.1097/00042737-200207000-00006. PMID 12169983
- [Background] Kohler N, Zeiser R. Intestinal Microbiota Influence Immune Tolerance Post Allogeneic Hematopoietic Cell Transplantation and Intestinal GVHD. Front Immunol. 2019 Jan 17;9:3179. doi: 10.3389/fimmu.2018.03179. eCollection 2018. PMID 30705680
- [Result] Ruckert T, Andrieux G, Boerries M, Hanke-Muller K, Woessner NM, Doetsch S, Schell C, Aumann K, Kolter J, Schmitt-Graeff A, Schiff M, Braun LM, Haring E, Kissel S, Siranosian BA, Bhatt AS, Nordkild P, Wehkamp J, Jensen BAH, Minguet S, Duyster J, Zeiser R, Kohler N. Human beta-defensin 2 ameliorates acute GVHD by limiting ileal neutrophil infiltration and restraining T cell receptor signaling. Sci Transl Med. 2022 Dec 21;14(676):eabp9675. doi: 10.1126/scitranslmed.abp9675. Epub 2022 Dec 21. PMID 36542690